CLINICAL TRIAL: NCT04893577
Title: A Randomized, Efficacy Assessor-Blinded, Study to Assess Preliminary Efficacy and Safety of EDTA Eye Drops v. an Active Comparator in the Suppression of Herpes Simplex Virus Eruptions in Subjects With a History of Herpes Labialis
Brief Title: EDTA Eye Drops Compared to Abreva for Herpes Simplex Virus Eruptions
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Christopher Hull, Assistant Professor, Dermatology, Principal Investigator, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB_00120663
Record Dates: First submitted 2021-05-14; First posted 2021-05-19 (Actual); Results first posted 2025-10-31 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Herpes Simplex Oral
MeSH Terms: conditions — Stomatitis, Herpetic | interventions — Edetic Acid; docosanol

STUDY DESIGN:
Intervention Model Description: This will be a randomized, efficacy assessor-blinded, parallel group, pilot study.
Who Masked: Outcomes Assessor
Masking Description: The subject and principal investigator will be unblinded, and only efficacy assessments will be done by a qualified trained blinded assessor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study Drug (EDTA Eye Drops) (Experimental): Patients will treat herpes simplex eruption with EDTA eye drops.
  Interventions: Drug: EDTA
- Active Comparator (Abreva) (Active Comparator): Patients will treat herpes simplex eruption with Abreva.
  Interventions: Drug: Abreva

INTERVENTIONS:
Drug: EDTA — Patients will treat their cold sore with EDTA eye drops based upon their randomization.
  Arms: Study Drug (EDTA Eye Drops)
Drug: Abreva — Patients will treat their cold sore with Abreva based upon their randomization
  Other Names: docosanol
  Arms: Active Comparator (Abreva)

SUMMARY:
This will be a randomized, efficacy assessor-blinded, parallel group, pilot study of up to 20 subjects with documented herpes labialis. Patients will be treated with the study drug, EDTA Eye Drops or the active comparator of Abreva.

Potential subjects will be assessed during a screening visit that must take place no greater than 2 weeks prior to the Day 1 (Baseline) visit. During the screening period, subjects that meet all other entry criteria will undergo UV susceptibility testing to determine their individual MED (minimal erythemal dose). UV susceptibility testing takes place over two days with exposure to UV light on specified regions on the subject's back followed by an assessment of the exposed areas 24 hours later to identify the MED. Subjects who have a measurable MED will be allowed to enroll in the study. Each subject will be randomly assigned in a 1:1 ratio to receive either EED or Comparator.

Patients who express a cold sore will track the lesion with a diary card to rate their pain levels, and any unusual symptoms at Day 1, Day 3, Day 5, Day 7, and Day 10. Patients may also take photographs of the lesion throughout the study.

DETAILED DESCRIPTION:
1.1 Background and Rationale Herpes simplex virus (HSV) infections are common and can cause significant morbidity both at the time of the original infection and when recurrences occur. There are two types of HSV - HSV-1 and HSV-2. HSV-1, the most common cause of oral "cold sores," is transmitted mainly by oral-to-oral contact. Genital herpes is usually caused by HSV-2, although HSV-1 can also cause genital breakouts. Both HSV-1 and HSV-2 infections are lifelong, with the virus living in the ganglia of nerves that supply the area of the original infection and recurring sporadically in the same area of that nerve's innervation. Most infections and recurrences are asymptomatic, but infectious viral shedding can occur. Patients who are not asymptomatic can develop prodromes of tingling, pain or paresthesia, and eventually blisters and ulcerations with pain. Healing generally occurs within 10 to 19 days after onset in primary infection or within 5 to 10 days in recurrent infection. Lesions usually heal completely, but recurrent lesions at the same site may cause atrophy and scarring.

According to WHO, in 2012 an estimated 3.7 billion people under age 50 (67%) had HSV-1 infection globally. Some patients have predictable outbreaks after exposure to noxious stimuli, such as sunlight fever, menstruation, or stress.

Researchers have found that calcium signaling is involved in the translocation of the virus from the ganglia to the eruption site. It has been found that an increase of calcium levels in the extracellular matrix will precipitate the calcium signaling events that are causal to the migration of the HSV virus from the proximal ganglia to the eruption site. (Hunsperger 2003, Cheshenko 2003) Further, Husperger found in her experiments (in vitro) that the chelation of calcium greatly reduced the reactivation of the HSV virus.

EDTA Eye Drops (EED), which consists of a calcium chelator and a permeation enhancer, could be one such intervention. Livionex has had some anecdotal evidence that this intervention could work at preventing an HSV eruption and post prodromal viral shedding.

IRB-approved clinical studies of HSV-1 have been performed in normal human volunteers with a history of HSV-1, who develop recurrences with prodromes after exposure to UV light. We will use this technique to induce recurrences in susceptible, HSV-1 infected individuals then treat with EED or Comparator 5 times daily.

Abreva has been chosen as the Comparator product in this study because it is approved by the FDA for treatment of HSV-related cold sores. Dosing 5 times/day has been selected as the dosing regimen because that is the dosing regimen approved for Abreva by FDA. The manufacturers of Abreva recommend that subjects not be treated for greater than 10 days. A maximum of 7 days treatment with study product has been chosen for this study.

Thus, treatment in both groups of subjects, will be 5 times daily and will last until healing of the lesion, or up to 7 days following the onset of the prodrome.

2. OBJECTIVE To collect preliminary efficacy and safety data on the use of EED in subjects with a history of herpes labialis, following UV Radiation

This will be a randomized, efficacy assessor-blinded, parallel group, pilot study of up to 20 subjects with documented herpes labialis.

Potential subjects will be assessed during a screening visit that must take place no greater than 2 weeks prior to the Baseline visit. During the screening period, subjects that meet all other entry criteria will undergo UV susceptibility testing to determine their individual MED (minimal erythemal dose). UV susceptibility testing takes place over two days with exposure to UV light on specified regions on the subject's back followed by an assessment of the exposed areas 24 hours later to identify the MED.

Subjects who have a measurable MED will be allowed to enroll in the study. Each subject will be randomly assigned in a 1:1 ratio to receive either EED or Comparator.

On Day 1, subjects will undergo UV radiation at a level 3 times their MED. The exposed area of the lip will be marked with indelible ink and a baseline photograph may be taken. (Specifics on the process for UV exposure will be explained in the study manual.) Subjects will be dispensed study medication and instructed how to apply it to the exposed area. Dosing of the study product will be done 5 times daily, beginning at the time that a subject first senses the start of the prodromal phase. The EED is a clear viscous eye drop, and the Comparator is a white cream substance. Therefore, the subject and principal investigator will be unblinded, and only efficacy assessments will be done by a qualified trained blinded assessor.

Subjects will be given a diary card to record their pain levels, progression of lesion development and any unusual symptoms (not normally seen with their outbreaks).

On Days 3,4, 5, and 6 the subject will follow up via virtual video call with blinded assessors during which the subject's diary card will be reviewed and compliance with dosing checked. Video calls will take place on weekedays. If however, Study Days 3-6 fall on a weekend day virtual video visits will not occur and subjects will be asked to upload photos to a secure, private MyChart account. If the subject has noted any unusual symptoms, these will be discussed with medical personnel to determine if a treatment emergent adverse event has occurred or, if the subject has not started treatment, whether their medical history should be updated. A photo will be taken of the irradiated area (as marked on Day 1) and the subject will be discharged and reminded to follow up on Day 7.

On Day 7 the subject will follow up via virtual video call for assessment of the irradiated area. Study staff will review the subject diary to determine if the subject is correctly noting the lesion stage and whether or not they have experienced a treatment emergent adverse event. If the subject has not experienced any prodromal symptoms or an outbreak of HSV by Day 7, they will be released from the study. All other subjects will be asked to upload a photo of the radiated area to their private individual Dropbox folder and asked to continue with dosing as instructed. They will be discharged from the clinic with a reminder to return on Day 10.

On Day 10, the subject will return to the clinic for assessment of the irradiated area. Study staff will review the subject diary to determine if the subject is correctly noting the lesion stage and whether they have experienced a treatment emergent adverse event. More study product will be dispensed as needed, a photo of the irradiated area will be taken, and the subject will be discharged with a reminder call the clinic and schedule an end of study (EOS) visit as soon as their lesion is healed or at 7 full days of treatment, whichever comes first. Study staff will ensure that the subject is seen within 24 hours of occurrence of either of these two milestones.

The EOS visit is expected to be the final study visit. A photo will be taken of the irradiated area, the diary card will be carefully reviewed and study product (including empty containers) will be collected. Subjects who developed a lesion that has not yet healed will be given the option to begin taking a prn medication that has been previously prescribed to treat an outbreak.

If an adverse event has occurred but has not resolved by the EOS visit, the subject will be contacted once weekly and status of the AE noted until such time as the event has resolved.

STUDY TREATMENT EDTA Eye Drops Livionex Inc. has agreed to supply EED. It consists of 2.6% EDTA plus a permeation enhancer (MSM). EED will be packaged in standard dropper bottles and labeled as containing 2.6% EDTA plus MSM as a surfactant.

Comparator: Abreva Abreva, manufactured by Avinir Pharmaceuticals, is an antiviral agent approved by the FDA for treatment of cold sores. It is packaged in tubes of 2g each.

ELIGIBILITY:
Inclusion Criteria

To be eligible for enrollment, a subject must meet the following criteria:

1. Understands the requirements of the study and provides written informed consent prior to undergoing any study-related procedures.
2. Subject is a male or female between the ages of 18-65 years old, inclusive.
3. Fitzpatrick skin type II or III.
4. History of at least one year of herpes labialis induced by UV exposure.
5. Able to recall exact location of most common or most recent outbreak.
6. History of at least 50% of cold sore outbreaks occurring with UV (sun) exposure.
7. At least 1 HSV-1 outbreak within the past 12 months.
8. Experiences prodromal symptoms before HSV-1 outbreaks.
9. Subject is willing and able to comply with protocol-specified dosing, visits to the clinic and tracking of pain.

Exclusion Criteria

Subjects will be excluded from the study if they meet any of the following criteria:

1. Outbreak <2 weeks prior to enrollment.
2. History of herpes simplex vaccine.
3. On antiviral suppression within the past 30 days.
4. Requires more than acetaminophen for pain from recurrent HSV outbreaks.
5. On any systemic or topical steroid, immune suppressant or chemotherapeutic agent within the past 30 days.
6. Use of tanning beds, history of sunburn, or beach vacation <2 weeks prior to enrollment.
7. History of photosensitivity, lupus erythematosus, or current use of photosensitizing medication.
8. Current immunosuppressed state due to underlying disease (i.e. HIV infection) concomitant treatment (i.e. chemotherapy).
9. Current upper respiratory tract infection or any active illness that could trigger cold sores or affect overall health of the patient or the assessment of the study agent.
10. Pregnant or intending to become pregnant during the study.
11. Abnormal skin conditions in the area of the recurrent HSV1 outbreaks.
12. Enrolled in another clinical trial within the past 30 days.
13. Previously treated with EED.
14. On any analgesics or NSAIDs that cannot be stopped during the study.
15. Alcohol or drug abuse.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-01-20 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2025-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher M Hull, M.D., Principal Investigator — University of Utah
Locations (1):
- University of Utah MidValley Dermatology, Murray, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cheshenko N, Trepanier JB, Gonzalez PA, Eugenin EA, Jacobs WR Jr, Herold BC. Herpes simplex virus type 2 glycoprotein H interacts with integrin alphavbeta3 to facilitate viral entry and calcium signaling in human genital tract epithelial cells. J Virol. 2014 Sep 1;88(17):10026-38. doi: 10.1128/JVI.00725-14. Epub 2014 Jun 18. PMID 24942591
- [Background] Evans TG, Bernstein DI, Raborn GW, Harmenberg J, Kowalski J, Spruance SL. Double-blind, randomized, placebo-controlled study of topical 5% acyclovir-1% hydrocortisone cream (ME-609) for treatment of UV radiation-induced herpes labialis. Antimicrob Agents Chemother. 2002 Jun;46(6):1870-4. doi: 10.1128/AAC.46.6.1870-1874.2002. PMID 12019102
- [Background] Hunsperger EA, Wilcox CL. Capsaicin-induced reactivation of latent herpes simplex virus type 1 in sensory neurons in culture. J Gen Virol. 2003 May;84(Pt 5):1071-1078. doi: 10.1099/vir.0.18828-0. PMID 12692270
- [Background] Jensen LA, Hoehns JD, Squires CL. Oral antivirals for the acute treatment of recurrent herpes labialis. Ann Pharmacother. 2004 Apr;38(4):705-9. doi: 10.1345/aph.1D285. Epub 2004 Feb 13. PMID 14966254
- [Background] Raborn GW, Grace MG. Recurrent herpes simplex labialis: selected therapeutic options. J Can Dent Assoc. 2003 Sep;69(8):498-503. PMID 12954137
- [Background] Spruance SL. The natural history of recurrent oral-facial herpes simplex virus infection. Semin Dermatol. 1992 Sep;11(3):200-6. PMID 1390034
- [Background] Spruance SL, Rowe NH, Raborn GW, Thibodeau EA, D'Ambrosio JA, Bernstein DI. Peroral famciclovir in the treatment of experimental ultraviolet radiation-induced herpes simplex labialis: A double-blind, dose-ranging, placebo-controlled, multicenter trial. J Infect Dis. 1999 Feb;179(2):303-10. doi: 10.1086/314605. PMID 9878012
- [Background] Spruance SL, McKeough MB. Combination treatment with famciclovir and a topical corticosteroid gel versus famciclovir alone for experimental ultraviolet radiation-induced herpes simplex labialis: a pilot study. J Infect Dis. 2000 Jun;181(6):1906-10. doi: 10.1086/315528. Epub 2000 May 31. PMID 10837169

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Study Drug (EDTA Eye Drops) | Active Comparator (Abreva)
Started | 5 | 5
Completed | 5 | 4
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Study Drug (EDTA Eye Drops) | Active Comparator (Abreva) | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 10
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 46 [29 to 62] | 36.2 [19 to 57] | 41.1 [19 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 4 | 2 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 5 | 10
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Duration (Days) of Herpes Labialis Outbreak Until Healed
Description: We will measure the number of days until lesion is healed from start of lesion to lesion resolved.
Time Frame: Up to 14 days per patient
Measure: Mean (Full Range); unit: days
Arm/Group | Study Drug (EDTA Eye Drops) | Active Comparator (Abreva)
Number analyzed (Participants) | 5 | 5
days | 10.6 [8 to 13] | 8.25 [3 to 14]

ADVERSE EVENTS:
Time Frame: Adverse events were collected over 12 days from beginning of randomization to end of study and 2 day follow-up call.
Arm/Group | Study Drug (EDTA Eye Drops) | Active Comparator (Abreva)
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 2/5 | 0/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Drug (EDTA Eye Drops) (N=5) | Active Comparator (Abreva) (N=5)
Burning during application of study drug (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) — Burning with medication application

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-10): https://cdn.clinicaltrials.gov/large-docs/77/NCT04893577/Prot_SAP_000.pdf